CLINICAL TRIAL: NCT00171691
Title: Safety of Diclofenac Sodium Gel in Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VOSG-PN-309
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis
Keywords: Knee osteoarthritis, Topical NSAID, Diclofenac sodium
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

INTERVENTIONS:
Drug: Diclofenac Topical Sodium Gel 1%

SUMMARY:
This study will test the efficacy and safety of topical Voltaren in the treatment of knee osteoarthritis.

ELIGIBILITY:
Key Inclusion criteria

• Osteoarthritis of the knee

Key Exclusion criteria

* Other rheumatic disease, such as rheumatoid arthritis
* Active gastrointestinal ulcer during the last year
* Known allergy to analgesic drugs

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2004-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events
Number of laboratory values outside pre-determined ranges at Months 1, 3, 6, 9 and 12

SECONDARY OUTCOMES:
Incidence of serious treatment-emergent adverse events
Number of patients who discontinued study medication due to a treatment-emergent adverse event
WOMAC pain, physical function and stiffness scores at Months 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Consumer Health Inc., Parsippany, New Jersey, United States

REFERENCES:
- [Derived] Peniston JH, Gold MS, Alwine LK. An open-label, long-term safety and tolerability trial of diclofenac sodium 1% gel in patients with knee osteoarthritis. Phys Sportsmed. 2011 Sep;39(3):31-8. doi: 10.3810/psm.2011.09.1918. PMID 22030938